CLINICAL TRIAL: NCT05181475
Title: A Clinical Study to Evaluate the Long-term Efficacy and Safety of Sodium Oligomannate Capsules (GV-971)
Brief Title: Long-term Efficacy and Safety Study of GV-971
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Green Valley (Shanghai) Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GV-971-PMS-B
Record Dates: First submitted 2021-12-02; First posted 2022-01-06 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — GV-971

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sodium Oligomannate Capsules (GV-971) (Experimental): The recommended dose regimen for subjects: GV-971 450 mg (3 capsules) per dose, bid, po. in morning and evening
  Interventions: Drug: Sodium Oligomannate Capsules (GV-971)

INTERVENTIONS:
Drug: Sodium Oligomannate Capsules (GV-971) — Sodium Oligomannate Capsules, each capsule contains 150 mg of sodium oligomannate. The recommended treatment is oral administration, 450 mg (3 capsules) per dose, bid, in morning and evening.

SUMMARY:
Sodium Oligomannate Capsules (GV-971) has been approved for treatment of mild to moderate Alzheimer's disease and improving the cognitive function of patients. This study plans to observe, in the clinical patients, the long-term efficacy and safety of GV-971, as well as the changes in blood and gut microbiota biomarkers after treatment, to validate the mechanism of action of GV-971, in order to better guide the rational use of drug in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 50 to 85 years (inclusive), with no restriction on gender;
2. Patients who met criteria for "probable AD" by National Institute on Aging and Alzheimer's Association (NIA-AA) diagnostic criteria;
3. Patients with mild to moderate AD as characterized by Mini-Mental State Examination (MMSE) scores between 11 and 26, inclusive;
4. Patients who have received at least primary education and have capacity to complete the measurement of cognition and other tests as specified in the protocol;
5. Patients receiving GV-971 treatment prescribed by clinicians;
6. Sign the informed consent form.

Exclusion Criteria:

1. Patients who have received GV-971 treatment within 6 months prior to screening;
2. Patients who may be allergic to Sodium Oligomannate Capsules as judged by the investigator;
3. Female participants who are pregnant or lactating;
4. Patients who cannot cooperate to complete the follow-up inquiries;
5. Any other diseases or conditions that are inappropriate to participate in this clinical trial in the opinion of the investigator.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Actual)
Dates: Start 2021-12-07 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the ADAS-cog/11 score | Baseline, 48 weeks
  Change from baseline in Alzheimer's Disease Assessments Scale - cognitive (ADAS-cog/11) scale total score. The total score of ADAS-cog/11 is 0-70, with higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Change from baseline in ADAS-Cog/11 score | Baseline, 96 weeks
  Change from baseline in Alzheimer's Disease Assessments Scale - cognitive (ADAS-cog/11) scale total score. The total score of ADAS-cog/11 is 0-70, with higher scores mean a worse outcome.
Change from baseline in MMSE score | Baseline, 48 weeks, 96 weeks
  Change from baseline in Mini Mental State Examination (MMSE) score. The total score of MMSE is 0-30, with higher scores mean a better outcome.
Change from baseline in ADCS-ADL score | Baseline, 48 weeks, 96 weeks
  Change from baseline in Alzheimer's Disease Cooperative Study - Activities of Daily Living; 23-item Scale (ACDS-ADL23) score. The total score of ADCS-ADL23 is 0-78, with higher scores mean a better outcome.
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 48 weeks, 96 weeks
  The incidence of adverse events and adverse reactions of vital signs, laboratory tests, electrocardiogram, and early withdrawal from the study in patients treated with GV-971.

CONTACTS AND LOCATIONS:
Locations (40):
- China (40):
  - Beijing Chao-Yang Hospital, Beijing, Beijing Municipality
  - Peking University Shougang Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Lanzhou University Second Hospital, Lanzhou, Gansu
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - The First People's Hospital of Foshan, Foshan, Guangdong
  - Nanfang Hospital, Guangzhou, Guangdong
  - The Affiliated Brain Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - The Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - No.6 HeBei Provincial People's Hospital, Baoding, Hebei
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - The First Hospital of Changsha, Changsha, Hunan
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Wuxi Mental Health Center, Wuxi, Jiangsu
  - Wuxi No.2 People's Hospital, Wuxi, Jiangsu
  - Northern Jiangsu People's Hospital, Yangzhou, Jiangsu
  - Affiliated Zhongshan Hospital of Dalian University, Dalian, Liaoning
  - The Second Hospital of Dalian Medical University, Dalian, Liaoning
  - Central Hospital Affiliated to Shandong First Medical University, Jinan, Shandong
  - The Second Hospital of Shandong University, Jinan, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Shanghai 6th People's Hospital, Shanghai, Shanghai Municipality
  - Shanghai East Hospital, Shanghai, Shanghai Municipality
  - Shanghai Mental Health Center, Shanghai, Shanghai Municipality
  - Tongren Hospital Shanghai Jiao Tong University School Of Medicine, Shanghai, Shanghai Municipality
  - Xinhua Hospital Affiliated To Shanghai Jiao tong University School of Medicine, Shanghai, Shanghai Municipality
  - Zhongshan Hospital, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - West China School of Medicine/West China Hospital of Sichuan University, Chengdu, Sichuan
  - Sir Run Run Shaw Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The Affiliated Hospital of Hangzhou Normal University, Hangzhou, Zhejiang
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Tongde Hospital of Zhejiang Province, Hangzhou, Zhejiang
  - Zhejiang Hospital, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang